CLINICAL TRIAL: NCT01008254
Title: Interdisciplinary Mobility Approach To Reduction Of Facility-Acquired Pressure Ulcers
Acronym: TEAM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Tracey L. Yap, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: #1007523
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Musical prompt (Experimental)
  Interventions: Behavioral: Musical prompt
- Delayed musical prompt (Active Comparator)
  Interventions: Behavioral: Delayed musical prompt
- No musical prompt (No Intervention)
  Interventions: Other: No musical prompt

INTERVENTIONS:
Behavioral: Musical prompt — Repositioning and mobility education program administered to all facility staff combined with tailored musical prompt reminder that played every two hours, every day, during a 12 hour period, for 12 months.
  Arms: Musical prompt
Behavioral: Delayed musical prompt — Repositioning and mobility education program administered to all facility staff combined with tailored musical prompt reminder that played every two hours, every day, during a 12 hour period, for 6 months.
  Arms: Delayed musical prompt
Other: No musical prompt — No intervention.
  Arms: No musical prompt

SUMMARY:
Musical reminder will raise compliance with mobility in the long-term care setting and reduce facility-acquired pressure ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Long-term care resident
* MDS qualified

Exclusion Criteria:

* Self pay long-term care residents

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Reduction of Facility Acquired Pressure Ulcers | 2 years

SECONDARY OUTCOMES:
Organizational Change | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tracey L Yap, RN, PhD, Principal Investigator — University of Cincinnati College of Nursing

REFERENCES:
- [Derived] Yap TL, Kennerly SM, Simmons MR, Buncher CR, Miller E, Kim J, Yap WY. Multidimensional team-based intervention using musical cues to reduce odds of facility-acquired pressure ulcers in long-term care: a paired randomized intervention study. J Am Geriatr Soc. 2013 Sep;61(9):1552-9. doi: 10.1111/jgs.12422. Epub 2013 Aug 26. PMID 24028358